CLINICAL TRIAL: NCT04658602
Title: Restoration of Permanent Molars Affected With Molar-incisor-hypomineralization (MIH) Among a Group of Egyptian Children Using Composite Restorations or Preformed Metal Crowns : Two-arm Randomized Controlled Trial (Part III)
Brief Title: Restoration of Permanent Molars Affected With (MIH) Using Composite Restorations or Preformed Metal Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nada Mahmoud Abd El-Azim Mohamed (Other)
Responsible Party: Sponsor-Investigator, Nada Mahmoud Abd El-Azim Mohamed, Doctor/Dentist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ttt of teeth with MIH part III
Record Dates: First submitted 2020-11-09; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: Parallel groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Quadruple ( Participant, Care Provider, Investigator, Outcomes Assessor ) Blinding to the child participants and legal guardian of each participating child, operator, outcome assessor and statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct composite restoration (Active Comparator): Bulk-fill composite (Filtek bulk flow, 3M Espe ) will be used and covered using a nanohybrid copmosite (filtek XT, 3M Espe )
  Interventions: Procedure: Preformed stainless steal crown cemented by glass ionomer lutting cement (Ketac cem,3M Espe)
- Preformed metal crowns (Active Comparator): Preformed stainless-steal crowns cemented by glass ionomer lutting cement (ketac cem. 3M Espe )
  Interventions: Procedure: Preformed stainless steal crown cemented by glass ionomer lutting cement (Ketac cem,3M Espe)

INTERVENTIONS:
Procedure: Preformed stainless steal crown cemented by glass ionomer lutting cement (Ketac cem,3M Espe) — Covering the affected molar with preformed metal crown cemented by glass ionomer lutting cement

SUMMARY:
The aim of this study is to compare clinical outcome of using direct esthetic composite restorations in managing MIH cases and the use of preformed metal crowns.

DETAILED DESCRIPTION:
Molar incisor hypomineralization can represent a serious and challenging clinical management problem. Children with MIH require higher levels of treatment needs and demonstrate considerable management problems.

For most severely affected MIH molars, direct esthetic restorative materials or preformed metal crowns will be the treatments to choose between. A number of aspects which could support decision-making, however, are not clearly demarcated. First and foremost, it is not clear if both treatments are similarly acceptable for patients and providers.

ELIGIBILITY:
Inclusion Criteria:

1. Children with MIH in one fully erupted molar or more.
2. Age ranging from 7-12 years.
3. cooperative children
4. Good general health.

Exclusion Criteria:

1. patients participating in other experiments.
2. Patients with parents planning to move away within the following year.
3. Patients with only mildly affected MIH molars that do not require extensive restorative treatment.
4. MIH-affected molars that have a very poor prognosis and require extraction.
5. First permanent molars that are affected with other developmental defects, such as hypoplasia, dental fluorosis or amelogenesis imperfecta.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pain after the restoration Binary (yes or no ) | 12 month
  Questionnaire

SECONDARY OUTCOMES:
Acceptability of the treatment Binary (yes or no ) | 12 month
  Questionnaire
Restoration quality score index | 12 month
  (FDI criteria: criterion marginal adaptation
Health-related quality of life changes by the therapies | 12 month
  Measured as difference in child perceptions Questionnaire CPQ 8-10/11-14)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alanzi A, Faridoun A, Kavvadia K, Ghanim A. 2018. Dentists' perception, knowledge, and clinical management of molar-incisor-hypomineralisation in kuwait: A cross-sectional study. BMC oral health. 18(1):34. Bakkal M, Abbasoglu Z, Kargul B. 2017. The effect of casein phosphopeptide-amorphous calcium phosphate on molar-incisor hypomineralisation: A pilot study. Oral health & preventive dentistry. 15(2):163-167. Baroni C, Marchionni S. 2011. Mih supplementation strategies: Prospective clinical and laboratory trial. Journal of dental research. 90(3):371-376. Bekes K, Heinzelmann K, Lettner S, Schaller HG. 2016. Efficacy of desensitizing products containing 8% arginine and calcium carbonate for hypersensitivity relief in mih-affected molars: An 8-week clinical study. Clinical oral investigations. Bekes K, Steffen R. 2016. Das würzburger mih - konzept: Teil 1. Der mih - treatment need index (mih - tni). Ein neuer index zur befunderhebung und therapieplanung bei patienten mit molaren - inzisiven hypomineralisation Oralprophylaxe & Kinderzahnheilkunde. 38(4):165-170. Briggs A, Sculpher M. 1997. Commentary: Markov models of medical prognosis. BMJ. 314 (7077):345-345.Briggs AH, O'Brien BJ, Blackhouse G. 2002. Thinking outside the box: Recent advances in the analysis and presentation of uncertainty in cost-effectiveness studies. Annual Review of Public Health. 23(1):377-401. Byford, S., Knapp, M., Greenshields, J., Byford, S., Knapp, M., Greenshields, J., et al (2003) Cost-effectiveness of brief cognitive behaviour therapy Cost-effectiveness of brief cognitive behaviour therapy versus treatment as usual in recurrent deliberate self- versus treatment as usual in recurrent deliberate selfharm: a rational decision making approach. harm: a rational decision making approach. Psychological Psychological MedicineMedicine, 33, 977 Cuzick J. 2005. Rank regression. Encyclopedia of biostatistics vol 6. Wiley and Sons. de Souza JF, Fragelli CB, Jeremias F, Paschoal MAB, Santos-Pinto L, de Cassia Loiola Cordeiro R. 2017. Eighteen-month clinical performance of composite resin restorations with two different adhesive systems for molars affected by molar incisor hypomineralization. Clinical oral investigations. 21(5):1725-1733. Dworkin SL. 2012. Sample size policy for qualitative studies using in-depth interviews. Archives of sexual behavior. 41(6):1319-1320. Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA. 2016. Consort 2010 statement: Extension to randomised pilot and feasibility trials. Bmj. 355:i5239 Elhennawy K, Jost-Brinkmann PG, Manton DJ, Paris S, Schwendicke F. 2017a. Managing molars with severe molar-incisor hypomineralization: A cost-effectiveness analysis within german healthcare. Journal of dentistry. 63:65-71. Elhennawy K, Manton DJ, Crombie F, Zaslansky P, Radlanski RJ, Jost-Brinkmann PG, Schwendicke F. 2017b. Structural, mechanical and chemical evaluation of molar-incisor hypomineralization-affected enamel: A systematic review. Archives of oral biology. 83:272-281. Elhennawy K, Schwendicke F. 2016. Managing molar-incisor hypomineralization: A systematic review. Journal of dentistry. 55:16-24. Foster Page LA, Thomson WM, Jokovic A, Locker D. 2005. Validation of the child perceptions questionnaire (cpq 11-14). Journal of dental research. 84(7):649-652. Fragelli CM, Souza JF, Jeremias F, Cordeiro Rde C, Santos-Pinto L. 2015. Molar incisor hypomineralization (mih): Conservative treatment management to restore affected teeth. Brazilian oral research. 29. Fragelli CMB, Souza JF, Bussaneli DG, Jeremias F, Santos-Pinto LD, Cordeiro RCL. 2017. Survival of sealants in molars affected by molar-incisor hypomineralization: 18-month follow-up. Brazilian oral research. 31:e30. Gaardmand E, Poulsen S, Haubek D. 2013. Pilot study of minimally invasive cast adhesive copings for early restoration of hypomineralised first permanent molars with post-eruptive breakdown. European archives of paediatric dentistry : official journal of the European Academy of Paediatric Dentistry. 14(1):35-39. Gambetta-Tessini K, Marino R, Ghanim A, Calache H, Manton DJ. 2016. Knowledge, experience and perceptions regarding molar-incisor hypomineralisation (mih) amongst australian and chilean public oral health care practitioners. BMC oral health. 16(1):75.